CLINICAL TRIAL: NCT02081781
Title: Case Control Study of the Factors That Affected the Outcome of Treatment of Congenital Nasolacrimal Duct Obstruction
Brief Title: The Factors That Affected the Outcome of Treatment of Congenital Nasolacrimal Duct Obstruction
Status: Completed | Type: Observational
Sponsor: Cathay General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CGH-P103002
Record Dates: First submitted 2014-03-05; First posted 2014-03-07 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-03

CONDITIONS: Congenital Nasolacrimal Duct Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Probing, topical anesthesia: Nasolacrimal duct obstruction (NLDO) is a quite common condition among the infants. An imperforate membrane at the distal end of the nasolacrimal duct is the main cause of occlusion. Children with the signs of NLDO presenting with epiphora and/or mucous discharge were included in this study. Intervention with probing under topical anesthesia was performed on the same surgeon. And success rate was evaluated.
  Interventions: Procedure: Probing

INTERVENTIONS:
Procedure: Probing — A punctal dilator was used for dilating the punctum. The nasolacrimal system was irrigated through either the lower or upper punctum with a hollow 23-gauge irrigating cannula attached to a syringe. A #0 (or #00) Bowman probe was passed through either the lower or upper canaliculus into the lacrimal sac and then directed downward through the nasolacrimal duct into nasal cavity. A "Hard" resistance could be felt as the probe touched the end of the nasolacrimal duct. A "Pop" tactile sensation might be noted while the probe passing through an obstruction at the valve of Hasner.

SUMMARY:
The purpose of this study was to investigate various potential factors that affected the outcome of treatment of congenital nasolacrimal duct obstruction.

DETAILED DESCRIPTION:
Congenital nasolacrimal duct obstruction is a common condition during the first few years of childhood. Most cases may resolve spontaneously, but the remaining children whose blockage does not resolve may require primary probing. Controversy remains regarding the optimal timing of the probing procedure. Another controversy is related to the setting of surgery. Therefore, we try to investigate the factors that affected the outcome of treatment of congenital nasolacrimal duct obstruction under the same surgical doctor during the past 13 years in our hospital.

ELIGIBILITY:
Inclusion Criteria:

* a history of tearing and/or mucopurulent discharge beginning during the first few weeks of life
* anatomical nasolacrimal duct obstruction

Exclusion Criteria:

* previous probing
* glaucoma
* trauma
* lid malpositions
* craniofacial anomalies
* congenital mucocele of the nasolacrimal sac

Ages: 1 Week to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2014-02; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
probing success: both anatomical patency of the duct and functional free of symptoms | one week

CONTACTS AND LOCATIONS:
Overall Officials: Chih Heng Hung, M.D., Principal Investigator — Department of Ophthalmology, Cathay General Hospital
Locations (1):
- Department of Ophthalmology, Cathay General Hospital, Taipei, Taiwan, Taiwan

REFERENCES:
- [Background] Pediatric Eye Disease Investigator Group; Repka MX, Chandler DL, Beck RW, Crouch ER 3rd, Donahue S, Holmes JM, Lee K, Melia M, Quinn GE, Sala NA, Schloff S, Silbert DI, Wallace DK. Primary treatment of nasolacrimal duct obstruction with probing in children younger than 4 years. Ophthalmology. 2008 Mar;115(3):577-584.e3. doi: 10.1016/j.ophtha.2007.07.030. Epub 2007 Nov 8. PMID 17996306
- [Background] Miller AM, Chandler DL, Repka MX, Hoover DL, Lee KA, Melia M, Rychwalski PJ, Silbert DI; Pediatric Eye Disease Investigator Group; Beck RW, Crouch ER 3rd, Donahue S, Holmes JM, Quinn GE, Sala NA, Schloff S, Wallace DK, Foster NC, Frick KD, Golden RP, Lambert SR, Tien DR, Weakley DR Jr. Office probing for treatment of nasolacrimal duct obstruction in infants. J AAPOS. 2014 Feb;18(1):26-30. doi: 10.1016/j.jaapos.2013.10.016. PMID 24568978